CLINICAL TRIAL: NCT00014469
Title: A Phase II Trial of IV Busulfan (Busulfex) and Melphalan as a Preparatory Regimen Prior to Allogeneic Bone Marrow Transplantation for the Treatment of Advanced and High Risk Hematologic Malignancies
Brief Title: Combination Chemotherapy Followed by Bone Marrow Transplantation in Treating Patients With Advanced Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-126; P30CA008748 (NIH); P01CA023766 (NIH); MSKCC-00126; NCI-H01-0070
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; acute undifferentiated leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; refractory cytopenia with multilineage dysplasia; juvenile myelomonocytic leukemia; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — Busulfan; Melphalan; Methotrexate; Tacrolimus

INTERVENTIONS:
Drug: busulfan
Drug: melphalan
Drug: methotrexate
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of busulfan and melphalan followed by donor bone marrow transplantation in treating patients who have advanced hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antileukemic potential of busulfan and melphalan prior to allogeneic bone marrow transplantation in patients with advanced or high-risk hematologic malignancy.
* Determine the incidence of transplantation-related morbidity and mortality in patients treated with this regimen.
* Determine the incidence of acute and chronic graft-versus-host disease in patients treated with this regimen.

OUTLINE: Patients receive cytoreductive chemotherapy comprising busulfan IV over 2 hours every 6 hours for a total of 16 doses on days -8 to -5 and melphalan IV over 30 minutes on days -4 to -2. Patients undergo T-cell replete allogeneic bone marrow transplantation on day 0. For graft-versus-host disease prophylaxis, patients receive tacrolimus IV continuously or every 12 hours beginning on day -1 and continuing for 50 days to 6 months followed by a taper. Once oral medications are tolerated, patients switch to oral tacrolimus every 12 hours. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

Patients are followed weekly through day 100, every 6 weeks for 3 months, every 3 months for 1 year, and then every 3-6 months for 6 months.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Infant leukemia
  * Acute lymphoblastic leukemia in 3rd or greater remission or relapse
  * Undifferentiated or biphenotypic leukemia in 2nd or greater remission or relapse
  * Juvenile chronic myelogenous leukemia (CML)
  * Acute myelogenous leukemia (AML) in 3rd or greater remission or relapse
  * Primary advanced myelodysplastic syndrome (MDS) excluding refractory anemia (RA) and RA with ringed sideroblasts
  * Therapy-related MDS of any stage or AML
  * CML in 2nd or greater chronic phase, accelerated, or blastic phase
  * Acute leukemia, CML, or MDS but unable to tolerate total body irradiation (TBI) due to potential neurotoxicity (prior TBI, prior local radiotherapy,or under 2 years of age)
* No active CNS disease
* Related or unrelated bone marrow donor matched at HLA-A, B, and DR beta 1

PATIENT CHARACTERISTICS:

Age:

* Under 60 (over 60 considered on case-by-case basis)

Performance status:

* Karnofsky 70-100%
* Lansky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* AST and ALT less than 2 times upper limit of normal
* Bilirubin less than 1.5 mg/dL unless liver is involved with disease

Renal:

* Creatinine normal
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Asymptomatic with no prior risk factors OR
* LVEF greater than 50% if symptomatic

Pulmonary:

* Asymptomatic with no prior risk factors OR
* Diffusion capacity greater than 50% predicted (corrected for hemoglobin) if symptomatic

Other:

* No active uncontrolled viral, bacterial, or fungal infection
* Not pregnant or nursing
* Negative pregnancy test
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 6 months since prior allogeneic or autologous stem cell transplantation

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trudy N. Small, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States